CLINICAL TRIAL: NCT00675545
Title: A Phase II Study of Docetaxel Plus Carboplatin in Chemonaive Hormone-Refractory Prostate Cancer (HRPC) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Dr. Alvin Wong, National University Hospital, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR01/30/06
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Hormone-Refractory Prostate Cancer
MeSH Terms: interventions — Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- docetaxel and prednisolone (Experimental): Patients in study will receive both chemotherapeutic agents on day 1 and day 8 of every 21-day cycle as described below:
  * Docetaxel 30 mg/m2 over 1 hour IV infusion, followed by
  * Carboplatin (AUC 2) over 1 hour IV infusion
  * Additonal medication required: IV Dexamethasone 10 mg followed by PO dexamethasone 4 mg 8 hourly x 4 doses, starting 12 hours after starting iv docetaxel.
  Interventions: Drug: Docetaxel, Carboplatin

INTERVENTIONS:
Drug: Docetaxel, Carboplatin — Docetaxel Form: A white, lyophilized powder in vials of 50, 150, and 450 mg each, which should be stored at room temperature in a light-protected area.
  Carboplatin Form: Taxotere is supplied as a sterile, non-aqueous, viscous solution with an accompanying sterile diluent (13% ethanol in water for injection). 20 and 80 mg strengths are available.
  Other Names: Carboplatin (Paraplatin); Docetaxel (Taxotere®)

SUMMARY:
The primary objective is to determine the efficacy of docetaxel plus carboplatin as first line treatment in patients with hormone refractory prostate cancer.

DETAILED DESCRIPTION:
Docetaxel-prednisolone is the current standard in HRPC, based on 2 large randomized trials showing improved survival compared to mitoxantrone-prednisolone. Carboplatin has activity in prostate cancer and the combination of Docetaxel-carboplatin is known to be synergistic and is used with good effect in many cancers. The advantage of using this combination in prostate cancer is suported by clinical data: high response rates of docetaxel-carboplatin-estramustine (with G-CSF support) in a phase II trial (Oh, Halabi, Kelly et al. Cancer. 2003 Dec 15;98(12):2592-8), and additional effect of this combination in prior taxane failures (Oh, George, Tay. Clin Prostate Cancer. 2005 Jun;4(1):61-4). Carboplatin itself has activity and theoretically could target the more hormone resistant clones or neuroendocrine components of the tumor.(Di Sant' Agnese. J Urol. 1994 Nov;152(5 Pt 2):1927-31.) We are studying the combination of docetaxel-carboplatin both given in a weekly, low-dose fashion, without estramustine and without G-CSF. This is expected to be an effective and tolerable treatment for HRPC patients. We will be documenting (to our knowledge) for the first time in this trial the efficacy of the combination given in this particular dose and schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate.
2. At the time of enrollment, patients must have evidence of metastatic disease, with either measurable disease per RECIST criteria or non- measurable disease (i.e. positive bones scan) and PSA > 5 ng/mm3.
3. Disease progression following androgen deprivation therapy.
4. Progression is defined according to the PSA Working Group criteria (see 6.1.3 and 6.3).
5. Serum testosterone levels < 50 ng/mm3 (unless surgically castrate). Patients must continue androgen deprivation with an LHRH analogue if they have not undergone orchiectomy.
6. No use of an antiandrogen for at least 4 weeks.
7. Have not been treated with chemotherapy before.
8. ECOG performance status of <= 2.
9. Laboratory criteria for entry:

   * White blood cell (WBC) => 3000/mm3
   * Platelets => 100,000/mm3
   * AST < 2.5 x upper limit of normal
   * Calculated CCT of => 40 ml/min
10. Signed informed consent form.
11. Age: 30 years old and above

Exclusion Criteria:

1. Significant peripheral neuropathy defined as grade 2 or higher.
2. Within 4 weeks since completing external beam radiotherapy or 8 weeks since completing radiopharmaceutical therapy (strontium, samarium).
3. Concomitant chemotherapy or investigational agents.

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
efficacy of docetaxel plus carboplatin | evaluated every 3 cycles (9 weeks)
  The primary endpoint of the study is best overall response (complete or partial response) obtained from measurable target lesion or PSA, as defined using the modified RECIST criteria.

SECONDARY OUTCOMES:
duration of response and toxicity profile of docetaxel and carboplatin. | during patient's treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alvin Wong, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213
- [Background] Oh WK, Halabi S, Kelly WK, Werner C, Godley PA, Vogelzang NJ, Small EJ; Cancer and Leukemia Group B 99813. A phase II study of estramustine, docetaxel, and carboplatin with granulocyte-colony-stimulating factor support in patients with hormone-refractory prostate carcinoma: Cancer and Leukemia Group B 99813. Cancer. 2003 Dec 15;98(12):2592-8. doi: 10.1002/cncr.11829. PMID 14669278